CLINICAL TRIAL: NCT04716738
Title: Sexual Dysfunction, Quality of Life and Visceral Hyperalgesia in Women With Irritable Bowel Syndrome
Brief Title: Visceral Sensitivity in Women With BS and Sexual Dysfunction
Acronym: IBS
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Hospital General de Mexico (Other Government)
Collaborators: Miguel Motola Kuba (Unknown); María de Fátima Higuera de la Tijera (Unknown); Yoshua Flores Bravo (Unknown)
Responsible Party: Principal Investigator, Santiago Camacho, Principal Investigator, Hospital General de Mexico
Other Study IDs: DI/19/107/03/080
Record Dates: First submitted 2021-01-14; First posted 2021-01-20 (Actual); Last update posted 2022-09-29 (Actual); Status verified 2022-09

CONDITIONS: Irritable Bowel Syndrome; Sexual Dysfunction
Keywords: Visceral sensitivity; Barostat; Quality of life; Irritable Bowel Syndrome; Sexual dysfunction; Biological marker
MeSH Terms: conditions — Irritable Bowel Syndrome; Sexual Dysfunction, Physiological

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Irritable Bowel Syndrome with Sexual Dysfunction: We use Rome IV criteria, scale bristol and the female sexual fuction to establish IBS and sexual dysfunction diagnosis, and SF-36 to determinated quality of life.
  Interventions: Diagnostic Test: Blood analyses and coprological
- Irritable Bowel Syndrome without Sexual Dysfunction: We use Rome IV criteria, scale bristol and the female sexual fuction to establish IBS and sexual dysfunction diagnosis, and SF-36 to determinated quality of life.
  Interventions: Diagnostic Test: Blood analyses and coprological

INTERVENTIONS:
Diagnostic Test: Blood analyses and coprological — We will take a blood and stool sample

SUMMARY:
This study aims to compare visceral rectal sensitivity and quality of life of 40 Irritable Bowel Syndrome women, with (20) and without sexual dysfunction (20). Both Irritable Bowel Syndrome (IBS) and sexual dysfunction (SD), decrease quality of life (QOL) separately, and only recently we have shown that quality of life decreases even more with both diseases. Thus, there is clinical evidence to search for a biological marker that explains this cumulative effect. Investigators will determine IBS using the Rome IV criteria, SD through the Female Sexual Function Index (FSFI) while and QOL through the Short Form-36 and the IBS-QOL. Visceral sensitivity will be evaluated by a barostat study: A small bag connected to a computer is placed in the rectum. This computer will insufflate air increasing the volume and simultaneously record the pressure inside the rectum; therefore investigators can simulate what happens when the stool reaches the rectum. The patient reports the first sensation, gas sensation, need to defecate and even pain. For patient protection the pressure will never exceed 50 mmHg and/or if any amount of pain is reported. To assess the effect of food on this visceral sensitivity, it is performed in 2 stages, fasting and 30 minutes after a standardized meal. The protocol will be carried out through 3 visits. First patients will be recruited; the diagnosis of IBS, SD, quality of life will be established and basic laboratory tests will be schedule before next visit. Second visit will be on day 7 of the menstrual cycle when investigators will carry out the barostat study and determination of blood´s sex hormones. The last visit is for the second barostat study on day 21 of the menstrual cycle with sex hormones measurement. This protocol will compare: Rectal pressure and volume for tone, first sensation, gas sensation, desire to defecate and pain, measure during fasting and postprandial periods in day 7 and 21 (estrogenic and progesterone phase) of the menstrual cycle. Other variables include (age, marital status, disease history, SF-36, IBS-QOL, etc.). This study aims to find a biological marker to explain the low QOL observed in daily clinical practice. This approach will allow us a more effective diagnosis and perhaps the creation of more effective therapeutic approaches to treat these patients. In the long term, we expect to establish the foundations of a patient-centered medicine with shared decision more effective in the gut brain axis disorders.

DETAILED DESCRIPTION:
Irritable bowel syndrome (IBS) is characterized by chronic abdominal pain related to alterations in defecation. Although the diagnostic criteria used in various consensuses may mask its true prevalence and incidence, it is known that it suffers between 5 and 15% of the population and it is more than two times more frequent in women. Only 10% of patients seek medical attention and even so it represents between 25 and 50% of gastroenterological visits in the United States. In Mexico the frequency is similar to that reported in the world.

IBS does not have a specific biological marker, but it is known that there are multiple factors involved in its pathophysiology. However, alterations in the gut-brain (GBA) are considered the main mechanism in the generation of symptoms.

The GBA regulates homeostatic functions through a set of organs that form a bidirectional network that links both elements. The neural portion includes peripheral elements (enteric nervous system, ENS), related elements (pairs of spinal and cranial nerves) and central (superior brain nuclei).

The ENS (neurons in the intestinal wall, epithelial and endocrine elements, associated neurotransmitters, and visceral smooth muscle) is the third division of the autonomic nervous system.

Once sensory information is captured in peripheral receptors, the information travels by intrinsic innervation to generate local reflexes in the viscera (absorption, secretion, motility and sensitivity) or by extrinsic innervations of the vagus nerve and thoracolumbar sympathetic afferent pathways towards the spinal medulla.

The main route of afferent activation is through the prevertebral ganglia that carry the signal to the dorsal horns of the spinal cord that travel through the lateral spinothalamic tract that, through the thalamus; activates cortical areas of pain somatic location and by limbic areas for emotional evaluation. These changes in the brain connectome are diverse and it is an area in development.

This complex GBA relationship in IBS patients includes differences in sex, comorbidities, and quality of life (QOL). These differences include the activation of estrogen receptors distributed along the visceral pain pathways (ENS, spinal cord and brain centers) as they modulate the opening of ion channels, regulate the tachykinin receptor NK1 and induce substance release. Additionally, estrogens modulate visceral information in the CNS. Elevated estrogen in the amygdale, increase the sensomotor response to rectal distention in oophorectomized rats. There are also studies that suggest that estrogens may alter the expression of specific pain receptors such as the glucocorticoid receptor and involve the opioid system. Changes have been observed in brain structure and functional connectivity in women, as well as other sexual factors. There are multiple overlaps with other functional digestive diseases, non-digestive diseases, and psychological and psychiatric disorders.

These complex connections make us see the IBS as a multisystemic disorder with alterations in QOL and other comorbidities, such as sexual dysfunction (SD). Since 1987 it has been shown that up to 83% of patients with IBS have SD. In 1993 it was recognized that sexual abuse may be related to IBS and that it alters the perception of pain. In 1998, SD was positively associated with the severity of gastrointestinal symptoms. Patients with IBS have a greater number of problems of physical and psychological abuse, the symptoms are aggravated with menstruation and are related to hormonal changes.

On the other hand, patients with IBS have shown visceral hypersensitivity. The best method to determine visceral mechanical sensitivity is the barostat. Recently, it has been shown that there is a relationship between the severity of symptoms, quality of life, psychological stress, colonic transit and visceral hypersensitivity in patients with IBS. Patients with IBS and a history of severe physical/sexual abuse have visceral hyposensitivity. IBS presents a higher frequency of SD, as well as a deteriorated QOL and visceral hypersensitivity.

No studies with barostat and determination of QOL have been conducted in the same population of patients with IBS and SD, comparing them with patients with IBS and without SD.

Establishing the relationship between QOL, SD and possible visceral hypersensitivity will make it possible to characterize this population and thus be able to establish new therapeutic strategies.

General hypothesis: Women with IBS and SD have greater visceral rectal hypersensitivity than those without SD.

Primary objective: To evaluate the pattern of rectal visceral sensitivity in patients with IBS and SD and compare it with patients with IBS without SD.

Secondary: To assess the QOL in patients with IBS with and without SD. Universe: Women with IBS with and without sexual dysfunction, who are cared for in the Gastroenterology service of the General Hospital of Mexico.

Sample. Group 1: Patients with IBS and sexual dysfunction (n = 20). Group 1: Patients with IBS without sexual dysfunction (n = 20). The assignment of patients with IBS to the study group with and without sexual dysfunction will be according to the consecutive order in which they present to their clinic visit and after determining the Global Assessment of the Female Sexual Function Index.

Sample Size. The relationship between sample size, power and detectable difference was investigated, based on a previous study that evaluated the pain threshold recorded with the barostat in a problem group and a control group. The analysis was carried out comparing the two means with the unpaired Student's t, with two tails and an alpha value of 0.05. The anticipated standard deviation for each group resulted from the average between the standard deviation of the problem group (8.3) with the control group (8.8), resulting in a value of 8.5. The difference between means of the control group (35.9) and the problem group (27.2), resulted in 8.7. With this data a sample size of 16 subjects per group was obtained with a statistical power of 80%. Twenty women will be recruited to prevent the probable loss of 20%.

Measurements. Rome IV. The Rome IV, 2016criteria specify that abdominal pain must have occurred at least in the last 6 months with a frequency of at least once a week in the last 3 months and be related with at least 2 of the following characteristics: (a) Related to defecation, (b) Associated with changes in the frequency of defecation and / or (c) Associated with changes in the appearance of stool. The subtypes (constipation, diarrhea, mixed or indeterminate) are determined with the Bristol scale. Its application does not require special permissions.

Sexual function questionnaire. (Female Sexual Function Index, FSFI). The female sexual function index that we will use has been widely used in the Mexican population.40-42 It has 19 questions that evaluate 6 domains: Desire, arousal, lubrication, orgasm, satisfaction, and pain. The higher the score, the better the function. The optimal cut-off point to determine whether or not there is sexual dysfunction has been determined at 24.95 (sensitivity 64.15% and specificity of 75.76%). Does not require application permits.

General quality of life questionnaire (Short Form 36, SF-36). The SF-36 questionnaire has been adapted to the Mexican population and consists of 36 questions that assess 8 domains: physical function, physical role, body pain, general health, vitality, role emotional and mental health. The studies published on the characteristics of the Spanish version of the SF-36 provide enough evidence on its reliability, validity and sensitivity. Does not require application permits.

Specific Quality of Life Questionnaire for Irritable Bowel Syndrome (IBS-QOL) Developed in 199545 it has been used and widely validated in the Mexican population. It consists of 34 questions on a Likert scale from 1 to 5. It measures: Dysphoria, interference with activity , body image, health concern, food avoidance, social reaction, sexual concern and social relationship. The total score and scores in each dimension are converted on a scale from 0 to 100. Higher values indicate a better health-related quality of life. This questionnaire is copyrighted in favor of the MAPI institute.

Barostat Visceral sensitivity will be evaluated using a rectal barostat. After an overnight fast, a warm water enema will be performed 60 to 120 minutes before the study. Subjects will be studied without sedation and in the left lateral decubitus position. A rectal barostat distention will be placed 5 cm above the anal margin. Before starting the distension test, the subject will be warned that a rectal stimulus will be applied without her knowledge and when the light is illuminated on the perception panel, she must indicate her degree of pain perception. Gradual isobaric distention will be performed with increases of 4 mmHg from IOP. Strains will be performed to a grade 5 sensation or up to 50 mmHg (maximum strain pressure) or at the request of the subject. Each distension will be 1 minute in duration, and a 1 minute rest period will be observed between each step. At each pressure step, the volume of the bag will be recorded to assess rectal compliance. After 45 seconds of each distension step the light on the perception panel will illuminate to request the degree of rectal sensation of the subject under study. The intensity of the sensation will be quantified according to the control panel with numerical scales: 0 no sensation; 1 first sensation; 2 sensation of gas; 3 sensation of defecation; 4 mild pain; 5 moderate pain and 6: severe pain. Between each distension the pressure will return to the internal operating pressure. After this first phase, previously standardized foods will be taken. The meal will consist of 831 kcal and will be made with potato (100 g), mayonnaise (20 g), ham (100 g), margarine (20 g) and pineapple juice (250 ml). Each subject will consume the food completely in a maximum of 15 minutes. Thirty minutes after finishing the food, the postprandial tone and MLA will be measured.

STATISTIC ANALYSIS Parametric data will be compared using Student's t test. Nonparametric data will be compared using the Mann-Whitney U test. Symptoms and percentages will be evaluated with Fisher's exact test or chi square. The associations between data will be analyzed with the Spearman and Pearson correlation tests. The data will express the mean ± standard deviation and in percentages. Alpha = 0.05.

ELIGIBILITY:
Inclusion Criteria:

1. -18 Years And Older,
2. -Meet The Diagnostic Criteria Of Roma Iv For Ibs ,
3. - Agreeing To Participate In The Study And Sign Informed Consent

Exclusion Criteria:

1. -Patient With Non-Ibs-Related Visceral Neuropathy
2. - Prokinetic And/Or Antidepressant Treatment Within 3 Months
3. - Patients With Gastrointestinal Or Ibs-Related Disease
4. - Patients With Severe Heart, Kidney And/Or Systemic Diseases
5. - Pregnant Or Nursing Patients

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women with irritable bowel syndrome with and without sexual dysfunction who are cared for in the gastroenterology service of the general hospital of Mexico.
Sampling Method: Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2023-02-01 (Estimated); Primary Completion 2023-10-30 (Estimated); Study Completion 2023-11-01 (Estimated)

PRIMARY OUTCOMES:
Change on barostat study during menstrual cycle | Second and third visit: Day 7 and day 21 of the menstrual cycle
  In this procedure, a small bag is placed in the rectum which is connected to a computer. This computer will insufflate air (in mL), measuring the pressure (in mmHg) inside the viscus (in this case the rectum) all time. With this system, a very precise feedback system is created allowing decrease or increase the pressure inside the rectum and thereby provoke the perception in the patient of different sensations. With the barostat we can simulate what happens when the stool reaches the rectum. Thus, the patient can report a first sensation, gas sensation, the need to defecate and even pain (mild, moderate or intense)

SECONDARY OUTCOMES:
General Quality of Life questionnaire (SF-36, Short Form-36) | Baseline
  This questionnaire consists of 36 questions that evaluate 8 domains (Items): physical function (10), physical role (4), body pain (2), general health (5), vitality (4), social function (2), role emotional (3) and mental health (5). Additionally, the SF-36 has a transition item that asks about the change in general health status compared to the previous year. Items are coded, aggregated and transformed on a scale from 0 (worst health status for that dimension) to 100 (best health status). Scores for the physical and emotional scale can also be calculated through an orthogonal approach
Specific Quality of Life questionnaire (IBS-QOL, Irritable Bowel Syndrome-Quality of Life) | Baseline
  This questionnaire consists of 34 questions on a Likert scale from 1 to 5. It measures a total score and 8 dimensions (items): Dysphoria (8), interference with activity (7), body image (4), concern for health ( 3), food avoidance (3), social reaction (4), sexual concern (2) and social relationship (3). The total score and the scores in each dimension are converted on a scale from 0 to 100. Higher values indicate a better health-related quality of life

CONTACTS AND LOCATIONS:
Overall Officials: Santiago Camacho, MD, MSc, Principal Investigator — 6761

REFERENCES:
- [Background] Alammar N, Stein E. Irritable Bowel Syndrome: What Treatments Really Work. Med Clin North Am. 2019 Jan;103(1):137-152. doi: 10.1016/j.mcna.2018.08.006. PMID 30466670
- [Background] Black CJ, Yiannakou Y, Houghton LA, Ford AC. Epidemiological, Clinical, and Psychological Characteristics of Individuals with Self-reported Irritable Bowel Syndrome Based on the Rome IV vs Rome III Criteria. Clin Gastroenterol Hepatol. 2020 Feb;18(2):392-398.e2. doi: 10.1016/j.cgh.2019.05.037. Epub 2019 May 31. PMID 31154027
- [Background] Defrees DN, Bailey J. Irritable Bowel Syndrome: Epidemiology, Pathophysiology, Diagnosis, and Treatment. Prim Care. 2017 Dec;44(4):655-671. doi: 10.1016/j.pop.2017.07.009. Epub 2017 Oct 5. PMID 29132527
- [Background] Van den Houte K, Carbone F, Pannemans J, Corsetti M, Fischler B, Piessevaux H, Tack J. Prevalence and impact of self-reported irritable bowel symptoms in the general population. United European Gastroenterol J. 2019 Mar;7(2):307-315. doi: 10.1177/2050640618821804. Epub 2018 Dec 22. PMID 31080615
- [Background] Sperber AD, Dumitrascu D, Fukudo S, Gerson C, Ghoshal UC, Gwee KA, Hungin APS, Kang JY, Minhu C, Schmulson M, Bolotin A, Friger M, Freud T, Whitehead W. The global prevalence of IBS in adults remains elusive due to the heterogeneity of studies: a Rome Foundation working team literature review. Gut. 2017 Jun;66(6):1075-1082. doi: 10.1136/gutjnl-2015-311240. Epub 2016 Jan 27. PMID 26818616
- [Background] Aziz I, Simrén M. Irritable Bowel Syndrome. In: Reference Module in Biomedical Sciences. Elsevier; 2019. Available at: https://www-sciencedirect-com.pbidi.unam.mx:2443/science/article/pii/B978012801238366018X [Accessed July 1, 2019].
- [Background] Singh R, Salem A, Nanavati J, Mullin GE. The Role of Diet in the Treatment of Irritable Bowel Syndrome: A Systematic Review. Gastroenterol Clin North Am. 2018 Mar;47(1):107-137. doi: 10.1016/j.gtc.2017.10.003. PMID 29413008
- [Background] Lazaridis N, Germanidis G. Current insights into the innate immune system dysfunction in irritable bowel syndrome. Ann Gastroenterol. 2018 Mar-Apr;31(2):171-187. doi: 10.20524/aog.2018.0229. Epub 2018 Jan 18. PMID 29507464
- [Background] Awad RA, Martin J, Guevara M, Ramos R, Noguera JL, Camacho S, Santiago R, Ramirez JL, Toriz A. Defaecography in patients with irritable bowel syndrome and healthy volunteers. Int J Colorectal Dis. 1997;12(2):91-4. doi: 10.1007/s003840050088. PMID 9189778
- [Background] Awad RA, Camacho S, Martin J, Rios N. Rectal sensation, pelvic floor function and symptom severity in Hispanic population with irritable bowel syndrome with constipation. Colorectal Dis. 2006 Jul;8(6):488-93. doi: 10.1111/j.1463-1318.2006.01038.x. PMID 16784468
- [Background] Chong PP, Chin VK, Looi CY, Wong WF, Madhavan P, Yong VC. The Microbiome and Irritable Bowel Syndrome - A Review on the Pathophysiology, Current Research and Future Therapy. Front Microbiol. 2019 Jun 10;10:1136. doi: 10.3389/fmicb.2019.01136. eCollection 2019. PMID 31244784
- [Background] Khlevner J, Park Y, Margolis KG. Brain-Gut Axis: Clinical Implications. Gastroenterol Clin North Am. 2018 Dec;47(4):727-739. doi: 10.1016/j.gtc.2018.07.002. Epub 2018 Sep 28. PMID 30337029
- [Background] Jahng J, Kim YS. Irritable Bowel Syndrome: Is It Really a Functional Disorder? A New Perspective on Alteration of Enteric Nervous System. J Neurogastroenterol Motil. 2016 Apr 30;22(2):163-5. doi: 10.5056/jnm16043. No abstract available. PMID 27032542
- [Background] Gulbransen BD. Do nerves make bowels irritable? Am J Physiol Gastrointest Liver Physiol. 2018 Jul 1;315(1):G126-G127. doi: 10.1152/ajpgi.00129.2018. Epub 2018 Apr 19. No abstract available. PMID 29672154
- [Background] Mayer EA, Labus J, Aziz Q, Tracey I, Kilpatrick L, Elsenbruch S, Schweinhardt P, Van Oudenhove L, Borsook D. Role of brain imaging in disorders of brain-gut interaction: a Rome Working Team Report. Gut. 2019 Sep;68(9):1701-1715. doi: 10.1136/gutjnl-2019-318308. Epub 2019 Jun 7. PMID 31175206
- [Background] Vanner S, Greenwood-Van Meerveld B, Mawe G, Shea-Donohue T, Verdu EF, Wood J, Grundy D. Fundamentals of Neurogastroenterology: Basic Science. Gastroenterology. 2016 Feb 18:S0016-5085(16)00184-0. doi: 10.1053/j.gastro.2016.02.018. Online ahead of print. PMID 27144618
- [Background] Walsh KT, Zemper AE. The Enteric Nervous System for Epithelial Researchers: Basic Anatomy, Techniques, and Interactions With the Epithelium. Cell Mol Gastroenterol Hepatol. 2019;8(3):369-378. doi: 10.1016/j.jcmgh.2019.05.003. Epub 2019 May 18. PMID 31108231
- [Background] Awad RA, Santillan MC, Camacho S, Blanco MG, Dominguez JC, Pacheco MR. Rectal hyposensitivity for non-noxious stimuli, postprandial hypersensitivity and its correlation with symptoms in complete spinal cord injury with neurogenic bowel dysfunction. Spinal Cord. 2013 Feb;51(2):94-8. doi: 10.1038/sc.2012.98. Epub 2012 Aug 28. PMID 22929208
- [Background] Grundy D. Neuroanatomy of visceral nociception: vagal and splanchnic afferent. Gut. 2002 Jul;51 Suppl 1(Suppl 1):i2-5. doi: 10.1136/gut.51.suppl_1.i2. PMID 12077054
- [Background] Jiang Y, Greenwood-Van Meerveld B, Johnson AC, Travagli RA. Role of estrogen and stress on the brain-gut axis. Am J Physiol Gastrointest Liver Physiol. 2019 Aug 1;317(2):G203-G209. doi: 10.1152/ajpgi.00144.2019. Epub 2019 Jun 26. PMID 31241977
- [Background] Bhatt RR, Gupta A, Labus JS, Zeltzer LK, Tsao JC, Shulman RJ, Tillisch K. Altered Brain Structure and Functional Connectivity and Its Relation to Pain Perception in Girls With Irritable Bowel Syndrome. Psychosom Med. 2019 Feb/Mar;81(2):146-154. doi: 10.1097/PSY.0000000000000655. PMID 30615602
- [Background] Kim YS, Kim N. Sex-Gender Differences in Irritable Bowel Syndrome. J Neurogastroenterol Motil. 2018 Oct 1;24(4):544-558. doi: 10.5056/jnm18082. PMID 30347934
- [Background] Camacho S, Bernal F, Abdo M, Awad RA. Endoscopic and symptoms analysis in Mexican patients with irritable Bowel syndrome, dyspepsia, and gastroesophageal reflux disease. An Acad Bras Cienc. 2010 Dec;82(4):953-62. doi: 10.1590/s0001-37652010000400018. PMID 21152770
- [Background] Keefer L, Palsson OS, Pandolfino JE. Best Practice Update: Incorporating Psychogastroenterology Into Management of Digestive Disorders. Gastroenterology. 2018 Apr;154(5):1249-1257. doi: 10.1053/j.gastro.2018.01.045. Epub 2018 Feb 1. PMID 29410117
- [Background] Windgassen S, Moss-Morris R, Everitt H, Sibelli A, Goldsmith K, Chalder T. Cognitive and Behavioral Differences Between Subtypes in Refractory Irritable Bowel Syndrome. Behav Ther. 2019 May;50(3):594-607. doi: 10.1016/j.beth.2018.09.006. Epub 2018 Sep 21. PMID 31030876
- [Background] Faresjo A, Walter S, Norlin AK, Faresjo T, Jones MP. Gastrointestinal symptoms - an illness burden that affects daily work in patients with IBS. Health Qual Life Outcomes. 2019 Jul 1;17(1):113. doi: 10.1186/s12955-019-1174-1. PMID 31262316
- [Background] Guthrie E, Creed FH, Whorwell PJ. Severe sexual dysfunction in women with the irritable bowel syndrome: comparison with inflammatory bowel disease and duodenal ulceration. Br Med J (Clin Res Ed). 1987 Sep 5;295(6598):577-8. doi: 10.1136/bmj.295.6598.577. No abstract available. PMID 3117237
- [Background] Walker EA, Katon WJ, Roy-Byrne PP, Jemelka RP, Russo J. Histories of sexual victimization in patients with irritable bowel syndrome or inflammatory bowel disease. Am J Psychiatry. 1993 Oct;150(10):1502-6. doi: 10.1176/ajp.150.10.1502. PMID 8379554
- [Background] Scarinci IC, McDonald-Haile J, Bradley LA, Richter JE. Altered pain perception and psychosocial features among women with gastrointestinal disorders and history of abuse: a preliminary model. Am J Med. 1994 Aug;97(2):108-18. doi: 10.1016/0002-9343(94)90020-5. PMID 8059776
- [Background] Fass R, Fullerton S, Naliboff B, Hirsh T, Mayer EA. Sexual dysfunction in patients with irritable bowel syndrome and non-ulcer dyspepsia. Digestion. 1998;59(1):79-85. doi: 10.1159/000007471. PMID 9468103
- [Background] Reilly J, Baker GA, Rhodes J, Salmon P. The association of sexual and physical abuse with somatization: characteristics of patients presenting with irritable bowel syndrome and non-epileptic attack disorder. Psychol Med. 1999 Mar;29(2):399-406. doi: 10.1017/s0033291798007892. PMID 10218930
- [Background] Heitkemper MM, Cain KC, Jarrett ME, Burr RL, Hertig V, Bond EF. Symptoms across the menstrual cycle in women with irritable bowel syndrome. Am J Gastroenterol. 2003 Feb;98(2):420-30. doi: 10.1111/j.1572-0241.2003.07233.x. PMID 12591063
- [Background] Mulak A, Tache Y, Larauche M. Sex hormones in the modulation of irritable bowel syndrome. World J Gastroenterol. 2014 Mar 14;20(10):2433-48. doi: 10.3748/wjg.v20.i10.2433. PMID 24627581
- [Background] Eugenio MD, Jun SE, Cain KC, Jarrett ME, Heitkemper MM. Comprehensive self-management reduces the negative impact of irritable bowel syndrome symptoms on sexual functioning. Dig Dis Sci. 2012 Jun;57(6):1636-46. doi: 10.1007/s10620-012-2047-1. PMID 22290342
- [Background] Keszthelyi D, Troost FJ, Masclee AA. Irritable bowel syndrome: methods, mechanisms, and pathophysiology. Methods to assess visceral hypersensitivity in irritable bowel syndrome. Am J Physiol Gastrointest Liver Physiol. 2012 Jul 15;303(2):G141-54. doi: 10.1152/ajpgi.00060.2012. Epub 2012 May 17. PMID 22595988
- [Background] Simren M, Tornblom H, Palsson OS, Van Oudenhove L, Whitehead WE, Tack J. Cumulative Effects of Psychologic Distress, Visceral Hypersensitivity, and Abnormal Transit on Patient-reported Outcomes in Irritable Bowel Syndrome. Gastroenterology. 2019 Aug;157(2):391-402.e2. doi: 10.1053/j.gastro.2019.04.019. Epub 2019 Apr 22. PMID 31022401
- [Background] Ringel Y, Whitehead WE, Toner BB, Diamant NE, Hu Y, Jia H, Bangdiwala SI, Drossman DA. Sexual and physical abuse are not associated with rectal hypersensitivity in patients with irritable bowel syndrome. Gut. 2004 Jun;53(6):838-42. doi: 10.1136/gut.2003.021725. PMID 15138210
- [Background] Mearin F, Lacy BE, Chang L, Chey WD, Lembo AJ, Simren M, Spiller R. Bowel Disorders. Gastroenterology. 2016 Feb 18:S0016-5085(16)00222-5. doi: 10.1053/j.gastro.2016.02.031. Online ahead of print. PMID 27144627
- [Background] Rosen R, Brown C, Heiman J, Leiblum S, Meston C, Shabsigh R, Ferguson D, D'Agostino R Jr. The Female Sexual Function Index (FSFI): a multidimensional self-report instrument for the assessment of female sexual function. J Sex Marital Ther. 2000 Apr-Jun;26(2):191-208. doi: 10.1080/009262300278597. PMID 10782451
- [Background] Moreno-Lozano M, Duran-Ortiz S, Perez-Zavala R, Quinzanos-Fresnedo J. Sociodemographic factors associated with sexual dysfunction in Mexican women with spinal cord injury. Spinal Cord. 2016 Sep;54(9):746-9. doi: 10.1038/sc.2016.19. Epub 2016 Feb 23. PMID 26902463
- [Background] Cortes-Flores AO, Vargas-Meza A, Morgan-Villela G, Jimenez-Tornero J, Del Valle CJZ, Solano-Genesta M, Miranda-Ackerman RC, Vazquez-Reyna I, Garcia-Gonzalez LA, Cervantes-Cardona GA, Cervantes-Guevara G, Fuentes-Orozco C, Gonzalez-Ojeda A. Sexuality Among Women Treated for Breast Cancer: A Survey of Three Surgical Procedures. Aesthetic Plast Surg. 2017 Dec;41(6):1275-1279. doi: 10.1007/s00266-017-0960-6. Epub 2017 Aug 25. PMID 28842752
- [Background] Carranza-Lira S, Nunez FDC. Sexual dysfunction prevalence in a group of pre- and postmenopausal Mexican women. Prz Menopauzalny. 2018 Mar;17(1):39-42. doi: 10.5114/pm.2018.74901. Epub 2018 Apr 11. PMID 29725284
- [Background] Ware JE Jr, Sherbourne CD. The MOS 36-item short-form health survey (SF-36). I. Conceptual framework and item selection. Med Care. 1992 Jun;30(6):473-83. PMID 1593914
- [Background] Duran-Arenas L, Gallegos-Carrillo K, Salinas-Escudero G, Martinez-Salgado H. [Towards a Mexican normative standard for measurement of the short format 36 health-related quality of life instrument]. Salud Publica Mex. 2004 Jul-Aug;46(4):306-15. doi: 10.1590/s0036-36342004000400005. Spanish. PMID 15468571
- [Background] Patrick DL, Drossman DA, Frederick IO, DiCesare J, Puder KL. Quality of life in persons with irritable bowel syndrome: development and validation of a new measure. Dig Dis Sci. 1998 Feb;43(2):400-11. doi: 10.1023/a:1018831127942. PMID 9512138
- [Background] Remes-Troche JM, Torres-Aguilera M, Montes-Martinez V, Jimenez-Garcia VA, Roesch-Dietlen F. Prevalence of irritable bowel syndrome in caregivers of patients with chronic diseases. Neurogastroenterol Motil. 2015 Jun;27(6):824-31. doi: 10.1111/nmo.12556. Epub 2015 Mar 29. PMID 25817438
- [Background] Hou X, Chen S, Zhang Y, Sha W, Yu X, Elsawah H, Afifi AF, El-Khayat HR, Nouh A, Hassan MF, Fatah AA, Rucker Joerg I, Sanchez Nunez JM, Osthoff Rueda R, Jurkowska G, Walczak M, Malecka-Panas E, Linke K, Hartleb M, Janssen-van Solingen G. Quality of life in patients with Irritable Bowel Syndrome (IBS), assessed using the IBS-Quality of Life (IBS-QOL) measure after 4 and 8 weeks of treatment with mebeverine hydrochloride or pinaverium bromide: results of an international prospective observational cohort study in Poland, Egypt, Mexico and China. Clin Drug Investig. 2014 Nov;34(11):783-93. doi: 10.1007/s40261-014-0233-y. PMID 25258162
- [Background] Schmulson M, Ortiz O, Mejia-Arangure JM, Hu YB, Morris C, Arcila D, Gutierrez-Reyes G, Bangdiwala S, Drossman DA. Further validation of the IBS-QOL: female Mexican IBS patients have poorer quality of life than females from North Carolina. Dig Dis Sci. 2007 Nov;52(11):2950-5. doi: 10.1007/s10620-006-9689-9. Epub 2007 Apr 6. PMID 17415635
- [Background] Abel JL, Carson RT, Andrae DA. The impact of treatment with eluxadoline on health-related quality of life among adult patients with irritable bowel syndrome with diarrhea. Qual Life Res. 2019 Feb;28(2):369-377. doi: 10.1007/s11136-018-2008-z. Epub 2018 Sep 28. PMID 30267294
- [Background] Awad RA, Camacho S, Flores F, Altamirano E, Garcia MA. Rectal tone and compliance affected in patients with fecal incontinence after fistulotomy. World J Gastroenterol. 2015 Apr 7;21(13):4000-5. doi: 10.3748/wjg.v21.i13.4000. PMID 25852287
- [Background] Awad RA, Camacho S. A randomized, double-blind, placebo-controlled trial of polyethylene glycol effects on fasting and postprandial rectal sensitivity and symptoms in hypersensitive constipation-predominant irritable bowel syndrome. Colorectal Dis. 2010 Nov;12(11):1131-8. doi: 10.1111/j.1463-1318.2009.01990.x. PMID 19575740
- [Background] Ballantyne A, Eriksson S. Research ethics revised: The new CIOMS guidelines and the World Medical Association Declaration of Helsinki in context. Bioethics. 2019 Mar;33(3):310-311. doi: 10.1111/bioe.12581. No abstract available. PMID 30884547
- [Background] International Committee of Medical Journal Editors. Uniform requirements for manuscripts submitted to biomedical journals (excerpts). J Am Coll Dent. 2014 Summer;81(3):23-30. PMID 25951680
- [Derived] Camacho S, Diaz A, Perez P, Batalla H, Flores Y, Altamirano E, Higuera-de la Tijera MF, Murguia D, Gomez-Laguna L. Sexual dysfunction worsens both the general and specific quality of life of women with irritable bowel syndrome. A cross-sectional study. BMC Womens Health. 2023 Mar 27;23(1):134. doi: 10.1186/s12905-023-02272-9. PMID 36973732